CLINICAL TRIAL: NCT06477549
Title: Randomized Trial of Benadamustine Versus Ruxolitinib With Fludarabine and Busulfan Conditioning in Recipients of Haploidentical Stem Cell Transplantation
Brief Title: BeFluBu vs FluBuRux Conditioning in Haploidentical HCT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, Ivan S Moiseev, Vice-director of RM Gorbacheva Research Institute, St. Petersburg State Pavlov Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14/24-n
Record Dates: First submitted 2024-06-21; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Biphenotypic Acute Leukemia; Lymphoblastic Lymphoma; Myeloproliferative Neoplasm; Myelodysplastic Syndromes
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Biphenotypic, Acute; Myeloproliferative Disorders; Myelodysplastic Syndromes | interventions — Bendamustine Hydrochloride; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FluBeBu conditioning (Experimental): Days -7 through -2: Fludarabine 30 mg/m2/day iv x 6 days; Days -7 through -6: Bendamustine 90 mg/m2 iv x 2 days; Days -5 through -3: Busulfan 1 mg/kg po qid x 3 days;Days +3 through +4: Cyclophosphamide 50 mg/kg iv x 2 days; Days +5 through +20: ruxolitinib 5 mg tid per os; Days +21 through 150: ruxolitinib 5 mg bid per os.
  Interventions: Drug: Bendamustine Hydrochloride
- FluBeRux conditioning (Active Comparator): Days -7 through -2: Fludarabine 30 mg/m2/day iv x 6 days; Days -7 through -2: ruxolitinib 5 mg tid per os; Days -5 through -3: Busulfan 1 mg/kg po qid x 3 days; Days +3 through +4: Cyclophosphamide 50 mg/kg iv x 2 days; Days +5 through +20: ruxolitinib 5 mg tid per os; Days +21 through 150: ruxolitinib 5 mg bid per os.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Bendamustine Hydrochloride — Days -7 through -6: Bendamustine 90 mg/m2 iv x 2 days
  Arms: FluBeBu conditioning
Drug: Ruxolitinib — Days -7 through -2: ruxolitinib 5 mg tid per os
  Arms: FluBeRux conditioning

SUMMARY:
Haploidentical hematopoietic stem cell transplantation irrespective of the conditioning intensity and graft-versus-host disease prophylaxis is associated with high frequency of primary and secondary graft failure. Different technologies of with replete or depleted graft are associated with 7-20% of graft failures in different diseases. Fludarabine and busulfan conditioning is the most commonly used approach for a variety of diseases. In two previously completed trials of addition of either bendamustine and ruxolitinib to conditioning we observed low rates of primary graft failure with both approaches. The study is the direct randomized comparisons of these two approaches with the primary aim of reducing composite events of primary graft failure, relapse and non-relapse mortality. The stratas for the study are Disease Risk Index (DRI) and the age of the haploidentical donor (<35 vs ≥35).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have an indication for allogeneic hematopoietic stem cell transplantation with myeloablative conditioning for malignant disease
* Diagnosis: acute myeloid leukemia, acute lymphoblastic leukemia, mixed lineage acute leukemia, lymphoblastic lymphoma, chronic myeloid leukemia, myelodysplastic syndromes, myeloprolipherative neoplasm
* Age ≥18
* Malignant disease in hematologic response: <5% of clonal blasts in the bone marrow and no clonal blasts in peripheral blood.
* Patients with 5-9/10 HLA-matched related donor available. The donor and recipient must be identical by the following genetic loci: HLA-A, HLA-B, HLA-Cw, HLA-DRB1, and HLA-DQB1.
* Peripheral blood stem cells or bone marrow as a graft source

Exclusion Criteria:

* Titer of anti-donor anti-HLA antibodies ≥ 5000 at the time of inclusion
* Moderate or severe cardiac disease: ejection fraction <50%, unstable angina, stable angina NYHA class III or IV, chronic heart failure NYHA class III or IV, Lawn grade V arrhythmia, myocardial infarction within 3 months before inclusion
* Stroke within 3 months of inclusion, unless related to the underlying malignancy
* Severe decrease in pulmonary function: FEV1 <50% or DLCO<50% of predicted or respiratory distress or need for oxygen support;
* Severe organ dysfunction: AST or ALT >5 upper normal limits, bilirubin >1.5 upper normal limits, creatinine >2 upper normal limits
* Creatinine clearance < 40 mL/min
* Uncontrolled bacterial or fungal infection at the time of enrollment defined by CRP> 70 mg/L
* Requirement for vasopressor support at the time of enrollment
* Karnofsky index <70%
* Pregnancy
* Somatic or psychiatric disorder making the patient unable to sign informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | 2 years
  Measure: Kaplan-Meier estimate of either relapse, primary or secondary graft failure or death from all causes

SECONDARY OUTCOMES:
Cumulative incidence of primary and secondary graft failure | 365 days
  Cumulative primary and secondary graft failure, competing risk is death and relapse
Incidence of HSCT-associated adverse events (safety and toxicity) | 125 days
  Toxicity assessment is based on presence of NCI CTC AE 5.0 event grades 3-5. Veno-occlusive disease incidence and severity assessment is based on EBMT criteria 2020. Transplant-associated microangiopathy incidence assessment is based on Harmonization criteria by Schoettler et al. All toxicity measurements will be aggregated as severity scores
Infectious complications, including analysis of severe bacterial, fungal and viral infections incidence | 100 days
  proportion of patients, requiring systemic treatment for bacterial, viral and fungal disease
Cumulative incidence of acute GVHD grade II-IV | 125 days
  Cumulative incidence of patients with acute GVHD II-IV grade, competing risk is death, relapse and primary graft failure
Incidence of moderate and severe chronic GVHD | 2 years
  Cumulative incidence of patients with moderate and severe chronic GVHD according to NIH 2015 criteria, competing risk is death, relapse and primary graft failure
Non-relapse mortality analysis | 2 years
  Cumulative incidence of patients with mortality without hematological relapse of malignancy
Overall survival analysis | 2 years
  Measure: Kaplan-Meier estimate of death from all causes
GVHD-relapse-free survival analysis | 2 years
  Measure: Kaplan-Meier estimate of death, acute GVHD grade III-IV, severe chronic GVHD or relapse
Relapse cumulative incidence analysis | 2 years
  Cumulative incidence of patients with relapse, competing risk is non-relapse mortality

CONTACTS AND LOCATIONS:
Locations (1):
- RM Gorbacheva Research Institute, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Yes
Written proposal to the department of scientific affairs of Pavlov University with a subsequent signed contract for research
Supporting Information: Study Protocol
Time Frame: After final study analysis availability for 15 years
Access Criteria: Written proposal to the department of scientific affairs of Pavlov University with a subsequent signed contract for research

REFERENCES:
- Available data/document: Study Protocol: Protocol version 1.0 — https://cloud.mail.ru/public/wQ1q/8amGwZdMb — Study protocol signed